CLINICAL TRIAL: NCT04754568
Title: Virtual Reality Instructional Design in Orthopedic Physical Therapy Education: A Randomized Controlled Trial Comparing the Effects of Virtual Reality With Role-Playing Learning
Brief Title: Virtual Reality Instructional Design in Orthopedic Physical Therapy Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shenandoah University (Other)
Responsible Party: Principal Investigator, Aaron Hartstein, Associate Professor, Shenandoah University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: USD Paper 3
Record Dates: First submitted 2021-02-08; First posted 2021-02-15 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Virtual Reality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality instructional design (Experimental): Completion of virtual reality simulation of an outpatient physical therapy evaluation.
  Interventions: Other: Virtual reality instructional design
- Role-playing instructional design (Active Comparator): Completion of traditional role-playing of a scripted outpatient physical therapy evaluation
  Interventions: Other: Role-playing instructional design

INTERVENTIONS:
Other: Virtual reality instructional design — 60 minute immersive VR experience with branching method information delivery, physical therapy assessment, and diagnosis.
  Arms: Virtual reality instructional design
Other: Role-playing instructional design — 60 minute traditional role-playing with standardized patient
  Arms: Role-playing instructional design

SUMMARY:
The objective of this study is to assess the effects of virtual reality instructional design on physical therapy students' clinical decision-making skills, as compared with a traditional method of instruction with the same content and duration of exposure.

DETAILED DESCRIPTION:
An online random number generator will be used to randomize students into one of two groups: virtual reality instruction or role-paying instruction. All students will complete self-reported measures of clinical decision-making and metacognitive awareness prior to receiving their allocated instruction. While completing allocated instruction (either virtual reality or role-playing), measures of diagnostic accuracy and diagnostic efficiency will be collected. Following virtual reality or role-playing instruction, all included subjects will complete post-test measures of clinical decision-making ,metacognitive awareness, and engagement. One week later, all included subjects will be assessed on a musculoskeletal objective structured clinical examination (mOSCE).

ELIGIBILITY:
Inclusion Criteria:

* Students enrolled in their first year of physical therapy school at SU

Exclusion Criteria:

* Students enrolled in their second or third year of physical therapy school at SU

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Change in clinical decision-making | pre- and post-instructional design (immediately after completing virtual reality or role-playing)
  The Clinical Decision-Making Tool (CDM-Tool), a Likert-style questionnaire with 12 items, scored on a four-point scale. A higher raw score indicates a higher level of perceived decision-making ability.

SECONDARY OUTCOMES:
Change in metacognitive awareness | pre and post-instructional design (immediately after completing virtual reality or role-playing)
  Metacognitive Awareness Inventory (MAI), a Likert-style questionnaire with 52-items, scored on a five-point scale. A higher raw score indicates a higher level of perceived metacognitive awareness.
Self-reported measure of engagement | Post-instruction (immediately after completing either virtual reality or role-playing experience)
  Six-item, five-point Likert-style instrument. A higher raw score indicates greater level of student engagement.
Objective Structured Clinical Examination (OSCE) | 1 week following allocated instruction (either virtual reality or role-playing)
  Practical examination with 2 cases, assessing a student's ability to generate hypotheses, perform tests or measures to rule-in or rule-out hypotheses, and deliver an appropriate intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Patti Berg-Poppe, PT, PhD, Study Chair — University of South Dakota
Locations (1):
- Shenandoah University, Winchester, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kleinert R, Heiermann N, Plum PS, Wahba R, Chang DH, Maus M, Chon SH, Hoelscher AH, Stippel DL. Web-Based Immersive Virtual Patient Simulators: Positive Effect on Clinical Reasoning in Medical Education. J Med Internet Res. 2015 Nov 17;17(11):e263. doi: 10.2196/jmir.5035. PMID 26577020
- [Background] Middeke A, Anders S, Schuelper M, Raupach T, Schuelper N. Training of clinical reasoning with a Serious Game versus small-group problem-based learning: A prospective study. PLoS One. 2018 Sep 11;13(9):e0203851. doi: 10.1371/journal.pone.0203851. eCollection 2018. PMID 30204773
- [Background] Middeke A, Anders S, Raupach T, Schuelper N. Transfer of Clinical Reasoning Trained With a Serious Game to Comparable Clinical Problems: A Prospective Randomized Study. Simul Healthc. 2020 Apr;15(2):75-81. doi: 10.1097/SIH.0000000000000407. PMID 32044851